CLINICAL TRIAL: NCT00567892
Title: Collaborative Tinnitus Research at Washington University
Acronym: CTRWU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Professor, Washington University School of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-0689; R01DC009095 (NIH)
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-10

CONDITIONS: Subjective Tinnitus
Keywords: tinnitus; subjective tinnitus; therapy; repetitive transcranial magnetic stimulation; clinical trial
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. rTMS (Experimental): Stimulation Settings:
  Frequency -- 1Hz on 330 sec (5 min 30 sec.) per train for the first 5 trains with the last train 350 sec. (5 min. 50 sec.) in duration Off -- 90 sec (1 min. 30 sec.) Intensity -- 110% of motor threshold Duration -- 42½ minutes (total 2000 pulses in 6 trains)
  Interventions: Device: rTMS
- 2. Sham rTMS (Sham Comparator): Sham rTMS appears identical to and mimics sounds and sensations of active magnet.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Stimulation Settings:
  Frequency -- 1Hz on 330 sec (5 min 30 sec.) per train for the first 5 trains with the last train 350 sec. (5 min. 50 sec.) in duration Off -- 90 sec (1 min. 30 sec.) Intensity -- 110% of motor threshold Duration -- 42½ minutes (total 2000 pulses in 6 trains)
  Other Names: Neuronetics 2100 device

SUMMARY:
The goal of this trial to see if repetitive transcranial magnetic stimulation (rTMS) to the hearing area of the brain can lessen the perception of tinnitus. rTMS uses a strong magnet and when placed against the scalp generates a small electrical field within the brain. Depending on the frequency of the stimulation, this electrical field can either decrease or increase the electrical excitability of the brain. In this study, low-frequency stimulation will be used, which is thought to decrease nerve activity. It is this electrical excitability of the brain that is thought to be responsible for tinnitus.

The hypothesis of this study is that rTMS can decrease the perception of tinnitus.

DETAILED DESCRIPTION:
This will be a cross-over randomized trial. The order of the treatments received will be randomly selected and the participant will not be told which treatment they are receiving. Subjects will fall into one of the four treatment groups described below:

1. 2 weeks of active rTMS treatment followed by washout and then by 2 weeks sham
2. 2 weeks of sham followed by washout and then 2 weeks of active rTMS treatment
3. 4 weeks of active rTMS treatment followed by washout and then 4 weeks of sham
4. 4 weeks of sham followed by washout and then 4 weeks of active rTMS treatment

For the washout period between the two interventions, we will plan a minimum of 2 weeks to avoid the problem of carryover effects. Prior to starting the next intervention after the washout period, we will re-assess subject's tinnitus severity. To ensure no carryover effect, the washout period will be extended for those subjects whose tinnitus severity, as defined by the THI, is more than 20 points different than their baseline THI score.

ELIGIBILITY:
On-line eligibility screening:

https://tinnitus.wustl.edu/

Inclusion Criteria:

* Men and women between the ages of 18 and 60 years.
* Subjective, unilateral or bilateral, non-pulsatile tinnitus of 6 month's duration or greater.
* Tinnitus Handicap Inventory (THI) score of 38 or greater.
* Subjects of child-bearing potential using an appropriate form of birth control acceptable to the research team and with a negative urine pregnancy test or undergone sterilization procedure.
* Able to give informed consent.
* Available for once daily therapy, during working hours, Mon.-Fri.
* English-speaking.

Exclusion Criteria:

* Patients experiencing tinnitus related to cochlear implantation, retrocochlear lesion, or other known anatomic/structural lesions of the ear and temporal bone.
* Patients with hyperacusis or misophonia (hyper-sensitivity to loud noises).
* History of seizures, history of loss of consciousness requiring medical care, any other CNS pathology that increases a subject's risk for treatment with rTMS.
* Patients with cardiac pacemakers, intracardiac lines, implanted medication pumps, implanted electrodes in the brain, other intracranial metal objects with the exception of dental fillings, or any other contraindication for MRI scan.
* Any contraindication for receiving FDG PET, as determined by established clinical criteria.
* Patients with an acute or chronic unstable medical condition which, in the opinion of the investigator, would require stabilization prior to initiation of magnetic stimulation.
* Patients with any active ear disease that, in the opinion of the PI, needs to be further evaluated.
* Patients with symptoms of depression as evidenced by a score of 14 or greater on the Beck Depression Inventory or, in the opinion of the psychiatric sub-investigator demonstrates active mood symptoms that meet DSM-IV-TR criteria for Major Depressive Disorder.
* Any psychiatric co-morbidity that, in the opinion of the psychiatric sub-investigator, may complicate the interpretation of study results.
* Pregnancy
* Currently breast-feeding
* Previous treatment with rTMS
* Patients with tinnitus related to Workman's Compensation claim or litigation-related event.
* Patients with a history of diabetes.
* Fasting glucose > 150mg/Dl.
* Patients taking any medication(s), in the opinion of the investigator, that is(are) deemed to be etiologically related to the development of tinnitus.
* Unable to elicit a motor threshold with rTMS.
* A Mini-Mental Status Exam score less than 27.
* Untreated or newly diagnosed hypertension, (systolic blood pressures above 140 mm or diastolic pressure above 90 mm).
* Patients with a history of claustrophobia.
* Inability to lay flat for 2 hours.
* Active alcohol and/or drug dependence or history of alcohol and/or ETOH dependence within the last year.
* Any medical condition that, in the opinion of the investigators, confounds study results or places the subject at greater risk.
* Unable to provide informed consent.
* Any exclusions from radiology screening for MRI or PET scanning.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, CPI, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Medical Center, St Louis, Missouri, United States

REFERENCES:
- [Result] Piccirillo JF, Garcia KS, Nicklaus J, Pierce K, Burton H, Vlassenko AG, Mintun M, Duddy D, Kallogjeri D, Spitznagel EL Jr. Low-frequency repetitive transcranial magnetic stimulation to the temporoparietal junction for tinnitus. Arch Otolaryngol Head Neck Surg. 2011 Mar;137(3):221-8. doi: 10.1001/archoto.2011.3. PMID 21422304
- [Result] Pierce KJ, Kallogjeri D, Piccirillo JF, Garcia KS, Nicklaus JE, Burton H. Effects of severe bothersome tinnitus on cognitive function measured with standardized tests. J Clin Exp Neuropsychol. 2012;34(2):126-34. doi: 10.1080/13803395.2011.623120. Epub 2011 Dec 14. PMID 22168528
- [Result] Burton H, Wineland A, Bhattacharya M, Nicklaus J, Garcia KS, Piccirillo JF. Altered networks in bothersome tinnitus: a functional connectivity study. BMC Neurosci. 2012 Jan 4;13:3. doi: 10.1186/1471-2202-13-3. PMID 22217183
- [Derived] Piccirillo JF, Kallogjeri D, Nicklaus J, Wineland A, Spitznagel EL Jr, Vlassenko AG, Benzinger T, Mathews J, Garcia KS. Low-frequency repetitive transcranial magnetic stimulation to the temporoparietal junction for tinnitus: four-week stimulation trial. JAMA Otolaryngol Head Neck Surg. 2013 Apr;139(4):388-95. doi: 10.1001/jamaoto.2013.233. PMID 23599075

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period: August, 2008 to June, 2010
Pre-assignment Details: Screen failure reasons included: Screening for clinical depression or other significant psychiatric conditions, history of significant head injury, inability to obtain motor threshold with repetitive transcranial magnetic stimulation (rTMS), MRI claustrophobia, and two patients elected not to participate.
Groups:
- Active Then Sham rTMS Treatment (2 Weeks): Active rTMS Treatment for 2 weeks followed by 2 weeks wash-out and then 2 weeks sham. Subjects who do not return to within 20 points of Baseline THI at the end of 2 weeks washout will have washout extended up to 2 additional 2-week washout-periods.At the end of 6 weeks total washout, if the subject's THI remains greater than 20 points difference from bsseline THI subject will be considered to have completed the study and will not complete the second cross study arm. Subject will go staight to end of study visit.
- Sham Then Active rTMS Treatment (2 Weeks): Sham treatment for 2 weeks followed by 2 weeks wash-out and then 2 weeks Active rTMS Treatment.Subjects who do not return to within 20 points of Baseline THI at the end of 2 weeks washout will have washout extended up to 2 additional 2-week washout-periods.At the end of 6 weeks total washout, if the subject's THI remains greater than 20 points difference from bsseline THI subject will be considered to have completed the study and will not complete the second cross study arm. Subject will go staight to end of study visit.
- Active Then Sham rTMS Treatment (4 Weeks): Active rTMS Treatment for 4 weeks followed by 2 weeks wash-out and then 4 weeks sham.Subjects who do not return to within 20 points of Baseline THI at the end of 2 weeks washout will have washout extended up to 2 additional 2-week washout-periods.At the end of 6 weeks total washout, if the subject's THI remains greater than 20 points difference from bsseline THI subject will be considered to have completed the study and will not complete the second cross study arm. Subject will go staight to end of study visit.One subject had a drop of THI larger than 20 points from baseline after first arm of treatment and did not get the second arm.
- Sham Then Active rTMS Treatment (4 Weeks): Sham treatment for 4 weeks followed by 2 weeks wash-out and then 4 weeks Active rTMS Treatment. Subjects who do not return to within 20 points of Baseline THI at the end of 2 weeks washout will have washout extended up to 2 additional 2-week washout-periods.At the end of 6 weeks total washout, if the subject's THI remains greater than 20 points difference from bsseline THI subject will be considered to have completed the study and will not complete the second cross study arm. Subject will go staight to end of study visit.
Period: First Treatment (2 or 4 Weeks)
Arm/Group | Active Then Sham rTMS Treatment (2 Weeks) | Sham Then Active rTMS Treatment (2 Weeks) | Active Then Sham rTMS Treatment (4 Weeks) | Sham Then Active rTMS Treatment (4 Weeks)
Started | 7 | 7 | 10 | 10
Completed | 7 | 7 | 9 | 6
Not Completed | 0 | 0 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 4
Period: Washout (2 Weeks)
Arm/Group | Active Then Sham rTMS Treatment (2 Weeks) | Sham Then Active rTMS Treatment (2 Weeks) | Active Then Sham rTMS Treatment (4 Weeks) | Sham Then Active rTMS Treatment (4 Weeks)
Started | 7 | 7 | 9 | 6
Completed | 7 | 7 | 9 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Second Treatment (2 or 4 Weeks)
Arm/Group | Active Then Sham rTMS Treatment (2 Weeks) | Sham Then Active rTMS Treatment (2 Weeks) | Active Then Sham rTMS Treatment (4 Weeks) | Sham Then Active rTMS Treatment (4 Weeks)
Started | 7 | 7 | 9 | 6
Completed | 7 | 7 | 9 | 5
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 2 Week Treatment: Treatment (either active rTMS or sham)for 2 weeks followed by 2 week wash-out then treatment (opposite of first assignment)for 2 weeks
- 4 Week Treatment: Treatment (either active rTMS or sham)for 4 weeks followed by 2 week wash-out then treatment (opposite of first assignment)for 4 weeks
- Total: Total of all reporting groups
Arm/Group | 2 Week Treatment | 4 Week Treatment | Total
Number analyzed (Participants) | 14 | 20 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 20 | 34
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 52 (5.1) [42 to 59] | 42 [22 to 59] | 50 [22 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  United States | 14 | 20 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in THI (Tinnitus Handicap Inventory)
Description: Tinnitus Handicap Inventory (THI) is a measure of bother from tinnitus. THI is measured as a score in a scale ranging from 0=No bother to 100=Extremely Bothered. THI score post active rTMS treatment minus THI score pre active rTMS treatment will provide the change in THI score due to active treatment. THI score post rTMS sham minus THI score pre rTMS sham will provide change in THI due to sham. The difference of THI change due to active treatment minus THI change due to sham will provide the THI change that is our primary outcome measure.
Time Frame: baseline at the start of each treatment period, end of each treatment period (2 or 4 weeks)
Population: Study participant that successfully completed both study parts active rTMS treatment and sham rTMS treatment were included in analysis.
Measure: Median (95% Confidence Interval); unit: units on a scale
Groups:
- 2-weeks rTMS Active Treatment: Daily rTMS for about 1 hour with active device settings (stimulation intensity at 110% of motor threshold), for 2 weeks.
- 2-Weeks Sham rTMS Treatment: Daily sham-rTMS for about 1 hour with sham device settings for 2 weeks.
- 4-weeks rTMS Active Treatment: Daily rTMS for about 1 hour with active device settings (stimulation intensity at 110% of motor threshold), for 4 weeks.
- 4-weeks rTMS Sham Treatment: Daily sham-rTMS for about 1 hour with sham device settings for 4 weeks.
Arm/Group | 2-weeks rTMS Active Treatment | 2-Weeks Sham rTMS Treatment | 4-weeks rTMS Active Treatment | 4-weeks rTMS Sham Treatment
Number analyzed (Participants) | 14 | 14 | 13 | 13
units on a scale | -5 [-14 to 0] | -6 [-12 to -2] | -10 [-12 to 3] | -6 [-12 to 4]
Statistical Analysis 1: Comparison: 2-weeks rTMS Active Treatment vs 2-Weeks Sham rTMS Treatment; The null hypothesis for this study was the difference between the change in THI score due to active rTMS treatment and the change in THI score due to rTMS sham was not different from 0; Test type: Superiority or Other; p = 0.944, Wilcoxon signed rank test — All statistical tests were two-sided and were evaluated at the α = 0.05 level of significance; Since the assumptions of parametric tests were not met we used non-parametric tests for the analysis; Median Difference (Net) = 0, 95% CI 2-sided [-6 to 4]
Statistical Analysis 2: Comparison: 4-weeks rTMS Active Treatment vs 4-weeks rTMS Sham Treatment; The null hypothesis for this study was the difference between the change in THI score due to 4 weeks active rTMS treatment and the change in THI score due to 4 weeks rTMS sham was not different from 0; Test type: Superiority or Other; p = 0.674, Wilcoxon signed rank test; The assumptions of parametric tests were not met; Median Difference (Net) = -4, 95% CI 2-sided [-9 to 10] — All statistical tests were two-sided and were evaluated at the α = 0.05 level of significance

2. Secondary Outcome: Perceived Global Impression of Change (PGIC: Number of Participants With Perceived Global Impression of Change (PGIC) of 1 or Greater
Description: PGIC is a 7 point scale ranging from -3 to +3,with 0 meaning no change,negative values reporting worsening of symptoms(Tinnitus), and values of +1 or above reporting perceived improvement of Tinnitus.
  PGIC score post active rTMS treatment treatment will provide subject's impression of change in tinnitue due to active treatment.PGIC score post rTMS sham will provide subject's impression of change in tinnitus due to sham. Number of subjects with scores of 1 or above are recorded to perceive improvement due to treatment of the corresponding study arm.
Time Frame: End of each treatment period (2 or 4 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- 2-Weeks Active rTMSTreatment: Daily rTMS for about 1 hour with active device settings (stimulation intensity at 110% of motor threshold)
- 2-Weeks Sham rTMS Treatment: Daily sham-rTMS for about 1 hour with sham device settings for 2 weeks).
- 4-Weeks Active rTMSTreatment: Daily rTMS for about 1 hour with active device settings (stimulation intensity at 110% of motor threshold), for 4 weeks.
- 4-Weeks Sham rTMS Treatment: Daily sham-rTMS for about 1 hour with sham device settings for 4 weeks.
Arm/Group | 2-Weeks Active rTMSTreatment | 2-Weeks Sham rTMS Treatment | 4-Weeks Active rTMSTreatment | 4-Weeks Sham rTMS Treatment
Number analyzed (Participants) | 14 | 14 | 13 | 13
participants | 1 | 3 | 3 | 5

ADVERSE EVENTS:
Time Frame: Up to 6 months.Minimum of 10 weeks in 2wk treatment, or 14 weeks in 4 week treatment.
Description: Subjects who had decrease in THI > 20 pts were followed for up to 6 months. All subjects were followed thru for 4 weeks post treatment.
Groups:
- 2 Weeks Treatment: Treatment (either active rTMS or sham) for two weeks followed by 2 weeks wash-out then treatment (opposite of first assignment)for two weeks
- Four Week Treatment: Treatment (either active rTMS or sham)for 4 weeks followed by 2 week wash-out then treatment (opposite of first assignment)for 4 weeks
Arm/Group | 2 Weeks Treatment | Four Week Treatment
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/20
Other Adverse Events (participants affected / at risk) | 7/14 | 3/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 2 Weeks Treatment (N=14) | Four Week Treatment (N=20)
Worsening of Tinnitus (Ear and labyrinth disorders) | 2 (4) | 1 (1) — Some reported worsening of tinnitus that was later followed by improvement of tinnitus. In all cases the worsening was temporary, no longer than a day or two.
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 1 (2) — One subject complained of ear pain, subject thought it was related to magnet placement.
Worsening of Menopausal Symptoms (Reproductive system and breast disorders) | 1/4 (10) | 0/7 (0) — 1 Subject complained of increased hot flashes and irritability for 10 days during treatment. Unsure if related to treatment.
Neck Stiffness or Pain (Musculoskeletal and connective tissue disorders) | 3 (7) | 1 (1)
Lightheaded feeling (Nervous system disorders) | 1 (2) | 0 (0) — One subject reported feeling lightheaded for a few minutes after treatment for 2 days of treatment. Resolved on its own each time, and did not continue.

LIMITATIONS AND CAVEATS:
Excluding subjects with Beck Depression Index of above 14 we treated an exclusive group of the Very bothered tinnitus patients, which may not be representative of the tinnitus population as a whole.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No